CLINICAL TRIAL: NCT05983198
Title: SatisfACtion: Phase I/II, Open-label, Multi-center Study of [225Ac]Ac-PSMA-R2 in Men With mHSPC and Heavily Pre-treated PSMA-positive mCRPC, With/Without Prior 177Lu-labelled PSMA-targeted Radioligand Therapy
Brief Title: Phase I/II Study of [225Ac]Ac-PSMA-R2 in PSMA-positive Prostate Cancer, With/Without Prior 177Lu-PSMA RLT
Acronym: SatisfACtion
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAAA802A12101; 2021-003478-30 (EudraCT Number)
Record Dates: First submitted 2023-07-24; First posted 2023-08-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: 225Ac-PSMA-R2; dose limiting toxicity; DLT; Escalation with Overdose Control; EWOC; pre- and post-177Lu-PSMA-RLT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group-1 (mCRPC/ post-177Lu) (Experimental): 1. Dose Escalation: All eligible participants with Metastatic Castration Resistant Prostate Cancer (mCRPC) who have received anti-cancer treatment (post-Androgen Receptor Pathway Inhibitors (ARPI), post-taxane based chemotherapy and heavily pre-treated and having already received prior 177Lu-labelled Prostate Specific Membrane Antigen (PSMA)-targeting Radioligand Therapy (RLT) will receive the starting dose of 7 Megabecquerel (MBq) of 225Ac-PSMA-R2 to determine the Maximum Tolerated Dose/Recommended Dose for Expansion (MTD/RDE) of Group 1.
  2. Dose Expansion: Once RDE is determined for Group 1, participants who have previously received 177Lu-PSMA-RLT will be enrolled in Group 1 dose expansion.
  Interventions: Drug: 225Ac-PSMA-R2; Radiation: 68Ga-PSMA-R2; Radiation: 68Ga-PSMA-11
- Group-2 (mCRPC/ pre-177Lu) (Experimental): 1. Dose Escalation: All eligible participants with mCRPC who have received anti-cancer treatment (post-Androgen Receptor Pathway Inhibitors (ARPI), prior taxane-based chemotherapy is not required, but have never been treated with 177Lu-labelled PSMA-targeted RLT (177Lu-labelled PSMA-targeted RLT treatment naïve) will receive the starting dose of 7 Megabecquerel (MBq) of 225Ac-PSMA-R2 to determine the Maximum Tolerated Dose/Recommended Dose for Expansion (MTD/RDE) of Group 2.
  2. Dose Expansion: Once RDE is determined for Group 2, participants naïve to 177Lu-labelled PSMA-targeted Radioligand Therapy (RLT) will be enrolled in Group 2 dose expansion.
  Interventions: Drug: 225Ac-PSMA-R2; Radiation: 68Ga-PSMA-R2; Radiation: 68Ga-PSMA-11
- Group 3 (mHSPC/ pre-177Lu) (Experimental): 1. Dose Escalation: All eligible participants with mHSPC (177Lu-labelled PSMA-targeted RLT treatment naïve), who are treatment naive or minimally treated with a) luteinizing hormone-releasing hormone (LHRH) agonist/antagonists or bilateral orchiectomy with or without first generation antiandrogen (e.g. bicalutamide, flutamide) b) CYP17 inhibitor or ARDT exposure. Patient in this group will start treatment with 225Ac-PSMA-R2 after group 1 and group 2 patients.
  2. Dose Expansion: Once RDE is determined for Group 3, participants will be enrolled in Group 3 dose expansion.
  Interventions: Drug: 225Ac-PSMA-R2; Radiation: 68Ga-PSMA-R2; Radiation: 68Ga-PSMA-11

INTERVENTIONS:
Drug: 225Ac-PSMA-R2 — PSMA-R2 is a ligand coupled with 225Ac an alpha emitting radionuclide
Radiation: 68Ga-PSMA-R2 — Kit for radiopharmaceutical preparation
Radiation: 68Ga-PSMA-11 — Kit for radiopharmaceutical preparation
  Other Names: Locametz

SUMMARY:
This is an open label, phase I/II, multi-center study in adult participants with metastatic hormone sensitive prostate cancer (mHSPC) and with metastatic castration resistant prostate cancer (mCRPC) who have received prior anti-cancer treatment and have a positive 68Ga-PSMA-11 PET scan. The purpose of this study is to learn if the study drug, [225Ac]Ac-PSMA-R2, is safe and tolerable, and has anti-tumor activity in treated patients.

Enrollment of all participants was not completed. The evaluated radioligand showed acceptable safety but limited benefit in metastatic prostate cancer

DETAILED DESCRIPTION:
The study contains three groups (Group 1, Group 2, and Group 3). Each group has a dose escalation part at a specific dosing schedule followed by a dose expansion part. The dose escalation parts in each group within each dosing schedule will establish the maximum tolerated dose or the recommended dose for expansion (MTDs/RDEs) of the 225Ac-PSMA-R2. Dose escalation decisions will be made by the Investigators and Novartis during dose escalation meetings (DEMs) based on safety and tolerability information. The dose expansion parts in each group group/dosing schedule will assess the anti-tumor activity in the mHSPC and mCRPC populations.

ELIGIBILITY:
Key Inclusion Criteria:

* Evidence of PSMA-positive disease by 68Ga-PSMA-11 PET/CT and eligible as determined by central reading
* Documented progressive mCRPC or mHSPC
* Adequate organ function
* Prior orchiectomy or ongoing ADT and should have received prior 177Lu-PSMA-RLT (Group1 dose escalation & expansion) or never received 177Lu-PSMA-RLT (Group 2 and Group 3 dose escalation & expansion).

Key Exclusion Criteria:

* Any other investigational agents within 28 days of the anticipated C1D1 of 225Ac-PSMA-R2 therapy
* Any systemic anti-cancer therapy within 28 days of the anticipated C1D1 of 225Ac-PSMA-R2 therapy
* Uncontrolled pain or incompatibility that may result in participant's lack of ability to comply with imaging procedures
* History of CNS metastases and symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression
* History of myocardial infarction, angina pectoris, or coronary artery bypass graft within 6 months prior to ICF signature and/or clinically active significant cardiac disease
* Diagnosis of other malignancies in the past three years expected to alter life expectancy or may interfere with disease assessment

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2029-11-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of DLTs during the DLT observation period | Up to 6 weeks after the first 225Ac-PSMA-R2 dose administration
  To determine the Recommended Dose for Expansion (RDE) and corresponding regimen for 225Ac-PSMA-R2 monotherapy in PSMA-positive in:
  * Group-1 (mCRPC): Participants previously treated with 177Lu-labelled PSMA-targeted RLT (post-177Lu).
  * Group-2 (mCRPC): Participants not treated previously with 177Lu-labelled PSMA-targeted RLT (pre-177Lu).
  * Group-3 (mHSPC): Participants not treated previously with 177Lu-labelled PSMA-targeted RLT (pre-177Lu).
Dose Escalation: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) by group and frequency schedule | From date of the first administration of 225Ac-PSMA-R2 till 30 days safety follow-up, assessed up to approximately 15 months
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Dose Escalation: Tolerability | Up to 6 weeks after the first 225AC-PSMA-R2 dose administration
  Frequency of dose interruptions, reductions, discontinuations, and dose intensity by group.
Dose Expansion: Overall Response Rate (ORR) | From date of the first administration of 225Ac-PSMA-R2 until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 15 months
  Overall Response Rate (ORR) is defined as the proportion of participants with confirmed best overall response (BOR) of complete response (CR) or partial response (PR) in soft tissue according to Prostate Cancer Working Group 3 (PCWG3) -modified RECIST v1.1 in absence of bone progression (as per PCWG3).

SECONDARY OUTCOMES:
Dose Escalation: Incidence and severity of AEs and serious adverse events (SAEs) | Up to 6 months after the last 225Ac-PSMA-R2 dose administration
  Analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Dose Expansion: Incidence and severity of AEs and serious adverse events (SAEs) | Assessed up to approximately 15 months.
  Analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Dose Escalation & Dose Expansion: Frequency of dose interruptions, reductions, discontinuations, and dose intensity by treatment. | At day 1 of each cycle (1 cycle = up to 6 weeks)
  Tolerability of study drug will be assessed by summarizing the number of and the reasons for dose delays and dose reductions. Dose intensity will also be tabulated by treatment group.
Dose Escalation: Overall Response Rate (ORR) | Assessed up to approximately 15 months.
  Overall Response Rate (ORR) is defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR) in soft tissue.
Dose Escalation & Dose Expansion: Disease Control Rate (DCR) | Assessed up to approximately 15 months.
  Disease control rate (DCR) is defined as the proportion of participants with confirmed best overall response (BOR) of complete response (CR), partial response (PR) or stable disease (SD).
Dose Escalation & Dose Expansion: Best Overall Response (BOR) | Assessed up to approximately 15 months.
  Best Overall Response (BOR) is defined as the best response recorded from the start of the treatment until disease progression.
Dose Escalation & Dose Expansion: radiographic Progression Free Survival (rPFS) | Assessed up to approximately 15 months.
  Radiographic progression free survival (rPFS) is defined as the time (in months) from the date of the first administration of 225Ac-PSMA-R2 to the date of radiographic progression as outlined in PCWG3 modified RECIST 1.1 or death due to any cause.
Dose Escalation & Dose Expansion: Overall Survival (OS) | Assessed up to approximately 15 months.
  Overall survival (OS) is defined as the time (in months) from the date of the first administration of 225Ac-PSMA-R2 to the date of death due to any cause.
Dose Escalation & Dose Expansion: Duration of Response (DoR) | Assessed up to approximately 15 months.
  Duration of response (DOR) is defined as the time (in months) from the date of the first documented response (CR or PR) to the date of first documented progression.
Dose Escalation & Dose Expansion: Time to first Symptomatic Skeletal Event (SSE) | Assessed up to approximately 15 months.
  Time to a first symptomatic skeletal event (SSE) is defined as the time (in months) from the first administration of 225Ac-PSMA-R2 to the date of SSE or death due to any cause.
Dose Escalation & Dose Expansion: Percentage of Participants with Biochemical Response by ALP and LDH | Assessed up to approximately 15 months.
  Biochemical responses by Alkaline Phosphatase (ALP) and Lactate Dehydrogenase (LDH) will be measured as best percentage change from baseline
Dose Escalation and Dose Expansion: Percentage of Participants with Biochemical Response by PSA | Assessed up to approximately 15 months.
  Biochemical responses as measured by Prostate Specific Antigen (PSA): PSA50 response is defined as the proportion of participants who have achieved ≥50% decrease from baseline at any time.
Dose Escalation and Dose Expansion: Pharmacokinetics characterization of 225Ac-PSMA-R2 | At Cycle (C) 1 Day (D) 1 at different measurement times, and one timepoint at C1 D2, C1 D3 and C1 D4
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization.
Dose escalation and dose expansion: To assess the impact of 225Ac-PSMA-R2 on participant reported outcomes | From baseline until 24 months after the end of treatment
  Change in heath related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (2):
  - BAMF Health, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
- Australia (2):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
- Novartis Investigative Site, Montreal, Quebec, Canada
- France (6):
  - Novartis Investigative Site, Dijon, Cote D Or
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No